CLINICAL TRIAL: NCT04040569
Title: A Phase I Dose Escalation Study of Single Fraction Pre-operative Partial Breast (S-PBI) for Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1183
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients in each dose cohort will be treated as a single group for dose escalation. The starting dose for the dose escalation portion will be 30 Gy. Subsequent cohorts of patients will receive an additional 4 Gy per treatment. If significant toxicity is encountered at the starting dose, a de-escalation will occur (step -1) to 26.5 Gy. As we are currently concluding an adjuvant single fraction phase I protocol (ClinicalTrials.gov Identifier: NCT02685332) to 30 Gy in a single fraction for early stage breast cancer, if we meet our endpoints of this study, we will start our dose escalation at 34Gy instead of the 30 Gy, as safety of the 30 Gy arm will have already been established.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-fraction stereotactic partial breast radiotherapy (Experimental): The primary objective is to escalate the dose of 1 fraction stereotactic partial breast radiotherapy utilizing the MR Linac,Gammapod or Cyberknife system to an ablative dose in the pre-operative setting to the primary tumor without exceeding the maximum tolerated dose in patients with early stage breast cancer.
  Interventions: Radiation: Radiomics on MRI

INTERVENTIONS:
Radiation: Radiomics on MRI — Through extracting and analyzing a large number of features from medical imaging, radiomics has shown promising results in treatment outcome prediction for many diseases including breast cancer (45-50). UTSW physics group has developed several new radiomic approaches and radiomic features, such as a multi-objective radiomics model(51) and a new radiomic "Shell" feature(52). As an exploratory end point for this trial, the investigators will explore the application radiomics using pre-treatment MRI, treatment parameters and clinical characteristics as input to predict pathological response of radiation therapy (XRT) based on pathology report of surgical tissues and local recurrence.

SUMMARY:
The purpose of this phase I trial is to evaluate dose-limiting toxicity while dose escalating single-fraction preoperative S-PBI to a presumed radioablative dose over 3 cohorts, starting with 30Gy in 1 fraction and advancing to 34Gy and 38Gy in 1 fraction.

DETAILED DESCRIPTION:
Preoperative stereotactic breast radiation may be beneficial as it offers the ability to target smaller treatment volumes than what has been achievable with adjuvant PBI (Nichols IJROBP 2010), track radiobiological response to radiation at time of surgical pathology, and allow the removal of all irradiated tissue to potentially minimize late effects.The purpose of this phase I trial is to evaluate dose-limiting toxicity while dose escalating single-fraction preoperative S-PBI to a presumed radioablative dose over 3 cohorts, starting with 30Gy in 1 fraction and advancing to 34Gy and 38Gy in 1 fraction. This would be accomplished on the CyberKnife or GammaPod. The GammaPod is a novel device dedicated to S-PBI utilizing a Cobalt-60 source (Yu Med Phys 2013), which offers a highly reproducible prone setup with a mean of 1.8mm of mismatch reported in 15 patients at the University of Maryland on consecutive scans (Yu JCO 2011). Implications of this research are far reaching, including determination of the maximally tolerated dose for preoperative S-PBI, pathologic complete response rates of early stage breast cancer to a predicted radioablative dose, radiographic markers of treatment response (radiomics), and translational research assessing mechanisms of immune and radiation response.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive epithelial (ductal, medullary, lobular, papillary, mucinous (colloid), or tubular) histologies of the breast 3 cm or less(T1-T2cN0) in women who have not undergone surgery or neoadjuvant endocrine or chemotherapy for current breast cancer diagnosis
2. Tumor must not involve the overlying skin based on imaging evaluation and/or clinical exam
3. Age >/= 18 years old and female
4. Greatest Tumor dimension is 3cm or less based on US. MRI measurements can be included only if performed BEFORE the biopsy
5. Tumor must be unifocal
6. The tumor must be visible on CT scan and/or preferably marked with clip(s) in tumor
7. Patients must undergo an MRI for work up to aid in tumor delineation and to rule out additional foci of disease. If additional foci of disease are present, they need to have a negative biopsy to proceed with treatment.If patient cannot have MRI, contrast enhanced digital mammography (CEDM) is allowed in place of MRI.
8. Clinically and radiographically node negative on ultrasound of the axilla or MRI
9. Estrogen receptor positive or Progesterone receptor positive and Her2neu negative
10. Ability to understand and the willingness to sign a written informed consent.
11. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to the start of study and for the duration of radiation therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months

Exclusion Criteria:

1. Multi-centric disease
2. Prior RT to the involved breast
3. Tumor size >3cm
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
5. Patients who are pregnant or lactating due to the potential exposure to the fetus to radiation therapy and unknown effects of radiation therapy to lactating females
6. Patients unable to have an MRI or contrast enhanced digital mammography (CEDM)
7. Prior ipsilateral breast cancer
8. Tumor less than 5mm from the skin surface on clinical exam and/or radiographic imaging
9. Patients with active Lupus or scleroderma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only study
Enrollment: 45 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Reach the maximum tolerated dose (MTD) | 5 years
  The primary objective is to escalate the dose of 1 fraction stereotactic partial breast radiotherapy utilizing the MR Linac, Gammapod or Cyberknife system to an ablative dose in the pre-operative setting to the primary tumor without exceeding the maximum tolerated dose in patients with early stage breast cancer. Done by escalating the dose of SBRT toward the tumorcidal dose of 38 Gy in fraction. Doses will be escalated an additional 3.5-4 Gy per treatment. The phase I portion of the study will be completed when either of the following events occur: 1) the MTD for a cohort is reached or 2) when delivery of a pre-determined highest dose of radiation (38 Gy) that has been deemed likely to be efficacious for treatment of early stage breast cancer is attained.Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Cosmesis outcome | 5 years
  Photographs of both breasts will be taken and cosmesis form will be graded by the patient and the radiation oncologist at twelve months from the start of therapy and at yearly intervals thereafter and an independent panel established at UTSW Medical Center will evaluate cosmesis at the end of study.
  Excellent: When compared to the untreated breast, there is minimal or no difference in the sizes, shape, or texture of the treated breast. There may be mild thickening or scar tissue within the breast or skin, but not enough to change the appearance Good: There is mild asymmetry in the size or shape of the treated breast as compared to the normal breast. The thickening or scar tissue within the breast causes only mild change in the shape Fair: There is obvious difference in the size and shape of the treated breast. This change involves ¼ or less of the breast Poor: Marked change in the appearance of the treated breast involving more than ¼ of breast tissue
Local Control | 5 years
  computed using Kaplan-Meier curves along with the 95% confidence interval
Acute Toxicity | 90 Days
  Exact binomial method will be used to calculate toxicity. Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Late Toxicity | 24 Months
  Exact binomial method will be used to calculate toxicity. Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.
Rates of Surgical Morbidity | 5 years
  Number of patients with surgical morbidity
Pathologic Complete Response Rates | 5 years
  Exact binomial method will be used to calculate the response rate.
Distant Disease-Free Survival | 5 years
  computed using Kaplan-Meier curves along with the 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahimi A, Leitch M, Dogan B, Liu Y, Alluri P, Arbab M, Li X, Parsons DDM, Kim DWN, Wandrey N, Farr D, Seiler S, Unni N, Nguyen A, Wooldridge R, Chiu TD, Lu W, Stojadinovic S, Visak J, Nwachukwu C, Patel I, Morgan H, Bahrami S, Stein M, McArthur HL, Sahoo S, Timmerman R. Ablative Preoperative Single-Fraction Radiation Dose Escalation Among Patients With Breast Cancer: A Phase 1 Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543689. doi: 10.1001/jamanetworkopen.2025.43689. PMID 41236737